CLINICAL TRIAL: NCT06735014
Title: Multicenter Longitudinal Imaging in ALS for Disease Biomarker Development
Brief Title: Multicenter ALS Imaging Study
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); Minnesota Office of Higher Education (Other Government)
Responsible Party: Sponsor
Other Study IDs: CMRR-2024-32796
Record Dates: First submitted 2024-11-22; First posted 2024-12-16 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: Magnetic Resonance Imaging; MRI; ALSFRS-R; ECAS; plasma neurofilament light; NfL
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with ALS: Adults with early stage ALS
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Plasma neurofilament light chain (NfL) quantification
- Participants without ALS: Control participants free from neurological disease
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Plasma neurofilament light chain (NfL) quantification

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Participants will undergo 3T MRI scanning of the brain and cervical spine MRIs
Diagnostic Test: Plasma neurofilament light chain (NfL) quantification — Participants will undergo a blood draw for the quantification of plasma neurofilament light chain

SUMMARY:
This is a multi-site study of ALS participants and healthy controls who will undergo brain and cervical spine MRIs and NfL blood testing at up-to 4 time points over the course of a year. The primary goal is to identify objective biomarkers of disease progression that are biologically relevant, linearly progressive, and sensitive to change.

DETAILED DESCRIPTION:
Recent developments in Magnetic Resonance Imaging (MRI), biophysical modeling, and computing have improved the sensitivity of imaging metrics to detect disease-related changes in the central nervous system in neurological disorders. This improved sensitivity has paved the way for utilizing these metrics as potential biomarkers of disease, in particular, to measure disease progression over short durations.

The investigators hypothesize that the multimodal analysis of MRI biomarkers (microstructure and morphology) from the brain and spine will improve sensitivity to detect disease-related changes over durations as short as 3 to 6 months. The hypothesis is based on prior work detecting longitudinal changes in brain microstructure over 6 months in an ALS cohort with modest change in functional measures over that time, and that a multimodal analysis combining brain and spine MRI measures can improve disease diagnosis accuracy.

In this project, the investigators will establish the scalability, sensitivity over shorter durations, and overall clinical trial readiness of these metrics through a three-site study. The investigators also propose to improve the sensitivity of imaging metrics by combining multiple complementary measures from the brain and spine in a longitudinal multimodal statistical framework. Additionally, the investigators will demonstrate how these imaging metrics correlate with fluid biomarkers and functional progression measures.

Upon completion of the project, the investigators anticipate that the enhanced sensitivity of our proposed longitudinal MRI biomarkers will have an impact on ALS treatment by providing novel surrogate markers as potential outcome measures for clinical trials. The expected increased effect size will also reduce the cohort size needed to conduct trials, thereby increasing their feasibility. Beyond the scope of clinical trials, these multimodal MRI biomarkers will serve as an objective measure of upper motor neuron degeneration at the single patient level. The MRI measures will also be cross validated with fluid biomarkers and will contribute to efforts to stratify ALS patients into clinically homogeneous cohorts.

Participants will be asked to complete 4 study visits over a 12-month period, with visits at baseline, 3 months, 6 months, and 12 months. Participants will receive an exam by a neurologist, blood draw, and MRI scan and will be asked to answer surveys about their medical history and ALS symptoms. Participants will be compensated for each visit via a prepaid card. Non-local participants living ≥100 miles from the research facility will be partially compensated for travel.

ELIGIBILITY:
For participants with ALS:

* < 36 months since onset of symptoms
* Definite, probable, lab supported-probable or possible ALS by El Escorial criteria OR definite, probable or possible ALS per Awaji-Shima Criteria
* Forced vital capacity within the last 90 days ≥ 60% of the predicted value
* Able to consent for themselves
* Able to read and speak English
* Clear of any contraindications for MRI

Exclusion Criteria:

* Individuals will be excluded if they have any condition that makes MRI unsafe or if they are unable to comply with instructions.
* All participants will undergo a neurologic examination at enrollment. Control participants with clinically significant abnormal findings on neurological examination will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with early-stage ALS
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Fiber Density | Baseline, 3 months, 6 months, 12 months
  This measure comes from the biophysical model used in brain imaging and is collected using MRI. It refers to the volume of the intra-axonal compartment per unit volume of the tissue. As this is a fraction it does not have a unit.
Fiber Cross-Section | Baseline, 3 months, 6 months, 12 months
  This measure comes from the biophysical model used in brain imaging and is collected using MRI. It refers to the change it fiber cross-section at the fiber bundle level when undergoing spatial normalization. This measure does not have a unit.
Orientation Dispersion | Baseline, 3 months, 6 months, 12 months
  This measure comes from the biophysical model used in brain imaging and is collected using MRI. Orientation dispersion is a measure of the uncertainty in the estimation of the fiber bundle orientation. It varies from 0 to 1 and does not have a unit. Higher values indicate greater uncertainty in estimation.
Intracellular Volume Fraction | Baseline, 3 months, 6 months, 12 months
  This measure comes from the biophysical model used in brain imaging and is collected using MRI. It is the proportion of the imaging voxel occupied by intracellular compartments. This ratio varies from 0 to 1 and does not have a unit. Larger values indicate greater density of intracellular compartments.
Free Water | Baseline, 3 months, 6 months, 12 months
  This measure comes from the biophysical model used in brain imaging and is collected using MRI. It represents the fractional volume of the free-water compartment. This is a ratio and it does not have a unit.
Cortical Thickness | Baseline, 3 months, 6 months, 12 months
  This measure is collected using MRI. It is the thickness of the cortical gray matter and is measured in millimeters.
Spinal Cord Cross-Sectional Area | Baseline, 3 months, 6 months, 12 months
  This measure is collected using MRI. It is the area of the spinal cord cross-section measured in millimeter square.
Spinal Cord Corticospinal Tract (CST) Fractional Anisotropy (FA) | Baseline, 3 months, 6 months, 12 months
  This measure is collected using MRI. It is a dimensionless scalar value between 0 and 1, indicating the degree of anisotropy (directionality) of water diffusion in the spinal cord's corticospinal tract. Higher values indicate higher anisotropy.

SECONDARY OUTCOMES:
Plasma neurofilament light (NfL) quantification | Baseline, 3 months, 6 months, 12 months
  Plasma NfL quantification will be reported in units of pg/ml.
ALS Functional Rating Scale, Revised (ALSFRS-R) | Baseline, 3 months, 6 months, 12 months
  The ALSFRS-R includes 12 questions. Each task is rated on a five-point scale from 0 (can't do) to 4 (normal ability). Individual item scores are summed to produce a reported score of between 0=worst and 48=best.
Edinburgh Cognitive and Behavioural Screen (ECAS) | At 3-month visit (optional)
  The ECAS is a 20-minute assessment of language, memory, verbal fluency, executive function, visuospatial function, and social cognition, which produce a number of subscales with a maximum total score of 136. Higher scores indicate better functioning.
Penn Upper Motor Neuron Score | Baseline
  The Penn Upper Motor Neuron Score (PUMNS) is a 28-item scale that measures upper motor neuron (UMN) signs in amyotrophic lateral sclerosis (ALS). The scale ranges from 0 (normal) to 32 (for widespread/severe UMN involvement) and evaluates the bulbar region (scores 0-4), upper limbs (scores 0-14), and lower limb (scores 0-14). Higher scores indicate greater disease burden.

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Pisharady, PhD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Northwestern University, Evanston, Illinois
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish deidentified and preprocessed data from this study through public neuroimaging repositories. To facilitate the reproduction of our findings, we will also publish the deidentified data used to produce the figures and tables in our publications. We will keep the names and other identifying information of participants confidential.